CLINICAL TRIAL: NCT06470711
Title: Mapping of Electrical Properties in the Brain.
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 24-003556; NCI-2024-04689 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-003556 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Malignant Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Participants complete a survey and undergo MRI on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates imaging methods for monitoring neural and electrical activity in the brain for improving clinical diagnosis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Optimize pulse sequence acquisitions for diffusion imaging on clinical MRI vendor systems.

II. Develop image-based MRI models (including diffusion-based MRI) that accurately depict the multi-regional electrical properties in the brain (e.g., resistivity, current) to inform of neural integrity and function (including white matter tract integrity) in diseased and non-diseased states.

III. Compare/correlate image-based MRI models (e.g., diffusion) with existing structural, physiologic, and functional MRI methods (e.g., tensor imaging, fMRI, DSC-MRI, etc).

IV. Further train image-based models/measurements with loco-regional benchmarks including (but not exclusive to) electrophysiologic monitoring, functional and structural tissue assays (from available biopsies), and correlative clinical features (e.g., histology, outcomes, treatment, etc).

OUTLINE: This is an observational study.

Participants complete a survey and undergo MRI on study.

ELIGIBILITY:
Inclusion Criteria:

* Aim 1: normal healthy volunteers
* Aim 2, 3, 4: participants included in IRB 16-002424, including those that have undergone surgical biopsy/resection for suspected or known glioma

Exclusion Criteria:

* Healthy volunteer unable to have an MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers and clinical neuro-oncology subjects with high grade glioma
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Identify diffusion MRI metrics [using conductivity tensor imaging (CTI)] that inform of regional electrical properties in the brain | Baseline
  At least 4 normal white matter regions of the brain will be analyzed. Fractional anisotropy (FA) and optimized diagnostic imaging (ODI) values will be compared to determine alignment within normal healthy white matter tracts (e.g. cortical spinal tract, corpus callosum).

CONTACTS AND LOCATIONS:
Overall Officials: Leland S. Hu, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials